CLINICAL TRIAL: NCT06985862
Title: Development of Artificial Intelligence Tools for the Detection of Stress Markers and Consideration of Stress States in the Monitoring of Subjects With Type 1 Diabetes
Acronym: SMART-T1D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-A02431-46
Record Dates: First submitted 2025-03-31; First posted 2025-05-22 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Type 1
Keywords: stress; voice markers; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Voice recording 4 days a day (Experimental): * Morning (first recording): Text reading (article 25.1 of the Declaration of Human Rights).
  * Noon (second recording): Counting from 1 to 20 at normal speed
  * Evening (third recording): Prolonged phonation of the vowel 'a' without catching your breath.
  * Bedtime (fourth recording): Free expression describing stressful moments of the day and their impact on diabetes management, for at least 30 seconds.
  Interventions: Other: Voice recording 4 times a day

INTERVENTIONS:
Other: Voice recording 4 times a day — * Morning (first recording): Text reading (article 25.1 of the Declaration of Human Rights).
  * Noon (second recording): Counting from 1 to 20 at normal speed
  * Evening (third recording): Prolonged phonation of the vowel 'a' without catching your breath.
  * Bedtime (fourth recording): Free expression describing stressful moments of the day and their impact on diabetes management, for at least 30 seconds.

SUMMARY:
Stress refers to all the reactions of an organism subjected to exogenous or endogenous stress. In the context of diabetes, stress plays a critical role. There are two forms of stress: acute and chronic, both of which can have a significant impact on patients' glycaemic control. Acute stress, if repeated, can cause rapid increases in blood glucose levels, while chronic stress can lead to insulin resistance. It is therefore essential to develop tools for recognising and quantifying stress states specific to patients with diabetes. These tools would provide a better understanding of the role of stress in diabetes management, paving the way for more targeted therapeutic interventions and improving patients' quality of life.

We are currently training algorithms using advanced machine learning and artificial intelligence techniques to recognise and quantify stress states using existing databases, including voice and physiological data. These technological advances will make it possible to identify moments of stress more accurately and provide appropriate responses, thereby contributing to better diabetes management.

The SMART-T1D study is an ancillary study of the EVASTRESS study.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has signed the SMART-T1D free and informed consent form
* Patient able to speak and read French

Exclusion Criteria:

* Mute patient.
* Patient with severe speech problems that may prevent voice recordings from being made.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Voice recording of participants | 14 days
  Daily voice recordings

SECONDARY OUTCOMES:
Diabetes-related distress in the test population | at inclusion and after 14 days
  DDS T1 is an indicator of overall diabetes distress (average of 17 items, rated 1 to 6 on a scale).
  A higher score indicates higher distress.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves Benhamou, Pr, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - CERITD (Centre d'Etudes et de Recherches pour l'Intensification du Traitement du Diabète), Évry
  - Grenoble University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: No